CLINICAL TRIAL: NCT00839358
Title: Midodrine and Albumin for Cirrhotic Patients in the Waiting List for Liver Transplantation
Brief Title: Effect of Midodrine and Albumine in the Prevention of Complications in Cirrhotic Patients Awaiting Liver Transplantation
Acronym: MACHT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Maternal-Infantil Vall d´Hebron Hospital (Other); Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Pere Gines, Chief of Hepatology Unit, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MACHT; 07/0443 (Other Grant/Funding Number: Fondo de Investigación Sanitaria); 07/90077 (Other Grant/Funding Number: Fondo de Investigación Sanitaria)
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Renal Failure; Hyponatremia; Sepsis; Hepatic Encephalopathy; Gastrointestinal Bleeding
Keywords: cirrhosis; renal failure; midodrine; albumine
MeSH Terms: conditions — Renal Insufficiency; Hyponatremia; Sepsis; Hepatic Encephalopathy; Gastrointestinal Hemorrhage; Fibrosis | interventions — Albumins; Midodrine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Albumin plus midodrine (Active Comparator): Albumin 40 g every 15 days during 1 year or until liver transplantation. Midodrine 5mg/8h. It can be increased according the value of mean arterial pressure. If there is no increase (defined as at least 10mmHGin MAP)midodrine can be increased at a dose of 10mg/8h. This treatment will be given during 1 year or until liver transplantation.
  Interventions: Drug: albumin; Drug: Midodrine
- salin solution plus pills (Placebo Comparator): Placebo of albumin in the same schedule thats in arm 1; placebo of midodrine in the same schedule thats in arm 1.
  Interventions: Drug: albumin; Drug: Placebo

INTERVENTIONS:
Drug: albumin — albumine 40 g every 15 days
  Other Names: Albumina Grifols
Drug: Midodrine — Midodrine 5mg/8 hs, can be increase up to 8mg/8hs if there is a lack of increase in at least 10mmHg in mean arterial pressure after 15 days of treatment.
  Other Names: Gutron
  Arms: Albumin plus midodrine
Drug: Placebo — saline solution
  Other Names: Grifols saline solution
  Arms: salin solution plus pills

SUMMARY:
The aim of this study is to evaluate the effect of prolonged administration of albumin and midodrine on the prevention of complications (renal failure, sepsis, hemorrhage, hepatic encephalopathy and hyponatremia) in patients with cirrhosis in the waiting list for liver transplantation. One hundred and ninety four patients with cirrhosis and awaiting a liver transplantation will include in the study. Patients will be randomized to receive albumin and midodrine (treatment group) or administration of placebo (saline for albumine) and tablets with excipients without midodrine (control group). Patients will be followed-up during 12th months. In the treatment group albumin will be given at a dose of 40g every 15 days and midodrine 5mg tid, in addition with lactitol (conventional doses) and the specific treatment that patients require by cirrhosis. The group control will receive placebo in the same way than the treatment group in addition with lactitol and the specific treatment that they require by their disease. In all the patients liver and renal function test, hormones determination (renin, aldosterone, noradrenaline), and cytokines will be determined in basal conditions. All these determinations will be repeated at month 1st,3rd, 6th and 12th months. Before the inclusion in the study neuropsychological test and critical flicker test will be performed to diagnose minimum EH. These tests will be repeated at 3rd, 6th and 12th months. All the determinations will be repeated at any time that the patients develop any complication considered as an end point. In baseline conditions and at 3rd and 6th months a questionnaire of quality of life (SF36) will be performed. During a year of follow-up the number of paracentesis that patients require, the incidence of renal failure and EH and their relationship with hormonal activity and cytokine levels, free transplant survival and quality of life will be recorded.

DETAILED DESCRIPTION:
End point: To evaluate the effect of long term administration of albumin and midodrine on the prevention of complications associated with cirrhosis in patients with cirrhosis awaiting for liver transplantation.

Secondary end points:

* To evaluate improvement in the ascites control
* To evaluate survival at 6 and 12 months.
* To evaluate the relationship between the development of complications and the activity of vasoconstrictor systems( renin, aldosterone and norepinephrine) as well as the levels of cytokines (TNF, IL6 and IL10)
* To evaluate quality of life
* To evaluate the presence and outcome of MHE

ELIGIBILITY:
Inclusion Criteria:

* Patients with cirrhosis in the waiting list for liver transplant
* Patients with ascites or diuretic treatment
* To have written inform consent

Exclusion Criteria:

* Systolic blood pressure ≥150 mmHg and or diastolic blood pressure≥90 mmHg
* To have been treated with transjugular intrahepatic portosystemic shunt (TIPS) or surgical shunts
* Antibiotic treatment in the previous week before the inclusion in the study
* Respiratory or cardiac failure
* HIV positive

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2008-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
To evaluate complications (renal failure, hepatic encephalopathy, hyponatremia, infection and gastrointestinal bleeding) in patients with cirrhosis awaiting for liver transplant. | When 97 patients are included (% of the whole population)

CONTACTS AND LOCATIONS:
Overall Officials: Pere Ginès, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic, Villarroel 170, Barcelona, Spain

REFERENCES:
- [Background] Alessandria C, Debernardi-Venon W, Carello M, Ceretto S, Rizzetto M, Marzano A. Midodrine in the prevention of hepatorenal syndrome type 2 recurrence: a case-control study. Dig Liver Dis. 2009 Apr;41(4):298-302. doi: 10.1016/j.dld.2008.09.014. Epub 2009 Jan 20. PMID 19158001
- [Background] Martin-Llahi M, Pepin MN, Guevara M, Diaz F, Torre A, Monescillo A, Soriano G, Terra C, Fabrega E, Arroyo V, Rodes J, Gines P; TAHRS Investigators. Terlipressin and albumin vs albumin in patients with cirrhosis and hepatorenal syndrome: a randomized study. Gastroenterology. 2008 May;134(5):1352-9. doi: 10.1053/j.gastro.2008.02.024. Epub 2008 Feb 14. PMID 18471512
- [Background] Wong F, Pantea L, Sniderman K. Midodrine, octreotide, albumin, and TIPS in selected patients with cirrhosis and type 1 hepatorenal syndrome. Hepatology. 2004 Jul;40(1):55-64. doi: 10.1002/hep.20262. PMID 15239086
- [Background] Salerno F, Gerbes A, Gines P, Wong F, Arroyo V. Diagnosis, prevention and treatment of hepatorenal syndrome in cirrhosis. Gut. 2007 Sep;56(9):1310-8. doi: 10.1136/gut.2006.107789. Epub 2007 Mar 27. No abstract available. PMID 17389705
- [Background] Guevara M, Gines P. Hepatorenal syndrome. Dig Dis. 2005;23(1):47-55. doi: 10.1159/000084725. PMID 15920325
- [Derived] Sola E, Sole C, Simon-Talero M, Martin-Llahi M, Castellote J, Garcia-Martinez R, Moreira R, Torrens M, Marquez F, Fabrellas N, de Prada G, Huelin P, Lopez Benaiges E, Ventura M, Manriquez M, Nazar A, Ariza X, Sune P, Graupera I, Pose E, Colmenero J, Pavesi M, Guevara M, Navasa M, Xiol X, Cordoba J, Vargas V, Gines P. Midodrine and albumin for prevention of complications in patients with cirrhosis awaiting liver transplantation. A randomized placebo-controlled trial. J Hepatol. 2018 Dec;69(6):1250-1259. doi: 10.1016/j.jhep.2018.08.006. Epub 2018 Aug 21. PMID 30138685